CLINICAL TRIAL: NCT00132327
Title: Analysis of Erythema Migrans Lesions
Brief Title: Analysis of Lyme Disease Lesions
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050219; 05-I-0219
Record Dates: First submitted 2005-08-18; First posted 2005-08-19 (Estimated); Last update posted 2018-12-03 (Actual); Status verified 2018-11-29

CONDITIONS: Erythema Migrans Lesions; Erythema Migrans
Keywords: Lyme Disease; Borrelia Burgdorferi; Inflammation; Skin; Host Response; Erythema Migrans Rash; Healthy Volunteer; HV
MeSH Terms: conditions — Glossitis, Benign Migratory; Lyme Disease; Inflammation

SUMMARY:
This study will analyze cells from erythema migrans lesions, the "bull's eye" rash of Lyme disease. Little is known about what happens in the skin when it is infected with Borrelia burgdorferi, the bacteria that cause Lyme disease. This study will examine and compare laboratory findings in skin biopsies from people with Lyme disease and from healthy normal volunteers to try to better understand the infection.

Healthy volunteers and people with untreated erythema migrans rash who are 18 years of age or older may be eligible for this study.

All participants undergo a clinical examination, blood tests, between two to four skin biopsies (removal of a small piece of tissue for laboratory examination), and complete two health questionnaires. The biopsies are taken from the erythema migrans lesion in patients with Lyme disease and from skin on the legs, forearms, buttocks, or side from healthy volunteers. To collect the tissue, the skin at the biopsy site is numbed with injection of a local anesthetic and a sharp instrument is then used to remove a round plug of skin about the size of a pencil eraser. The wound may be closed with one or two sutures, or allowed to heal without sutures. The sutures are removed after a week to 10 days.

Patients with Lyme disease receive treatment for their condition. In addition, at the time the sutures are removed and at 4 weeks, 6 months, and 12 months after their first visit they fill out a questionnaire and have additional blood tests.

DETAILED DESCRIPTION:
Little is known of the host and the bacteria response in vivo in patients with Lyme disease. In an attempt to better understand the pathology of erythema migrans (EM), we will use a variety of techniques to characterize patterns in skin biopsies from individuals with a diagnosis of EM and compared those to the patterns seen in biopsies from unaffected individuals. Biopsies from patients may also be evaluated for B. burgdorferi. Patients diagnosed with erythema migrans will have between 2 and 4 punch skin biopsies of affected area, and will return for 4 follow up visits in the course of a year. Therapy for Lyme disease will be offered. Healthy volunteers will have a screening visit, a visit for the skin biopsies and a follow up visit. Patients and healthy volunteers will be compensated for their time and inconvenience.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients:

Age greater than or equal to 18 years

Diagnosis of EM - an expanding annular lesion, at least 5 cm in diameter on a person with a history of exposure to the disease.

Exposure is defined as having been (less than or equal to 30 days before onset of EM) in wooded, brushy, or grassy areas (i.e., potential tick habitats) in an area in which Lyme disease is endemic.

A history of tick bite is not required.

The area of the erythema migrans lesion is suitable for biopsy. This excludes biopsies on the face, neck, scalp, and over the tibia.

Not know to be positive for RPR, HIV, HBsAg or HCV

Able to give consent

Healthy Volunteers:

Age greater than or equal to 18 years

Not positive for RPR, HIV, HBsAg or HCV.

Able to give consent

EXCLUSION CRITERIA:

Patients:

Antibiotic therapy for the current episode of Lyme disease

Oral corticosteroids within the past 2 weeks

History of severe skin disease (such as psoriasis, atopic dermatitis) in the last year.

Diagnosis of diabetes, active cancer, or autoimmune diseases.

Investigational drugs in the past month

History of forming large thick scars after skin injuries or surgery

History of excessive bleeding after cuts or procedures or on anticoagulation.

Use of steroid cream/ointment at the rash.

Healthy Volunteers:

History of Lyme disease, or serological evidence for Lyme disease

No oral corticosteroids within the past 2 weeks

History of severe skin disease (such as psoriasis, atopic dermatitis) in the last year.

Diagnosis of diabetes, cancer, autoimmune diseases.

Investigational drugs in the past month

History of forming large thick scars after skin injuries or surgery

No history of excessive bleeding after cuts or procedures or on anticoagulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2005-08-17; Study Completion 2018-11-29

CONTACTS AND LOCATIONS:
Overall Officials: Adriana R Marques, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). Lyme disease--United States, 2001-2002. MMWR Morb Mortal Wkly Rep. 2004 May 7;53(17):365-9. PMID 15129194
- [Background] Fraser CM, Casjens S, Huang WM, Sutton GG, Clayton R, Lathigra R, White O, Ketchum KA, Dodson R, Hickey EK, Gwinn M, Dougherty B, Tomb JF, Fleischmann RD, Richardson D, Peterson J, Kerlavage AR, Quackenbush J, Salzberg S, Hanson M, van Vugt R, Palmer N, Adams MD, Gocayne J, Weidman J, Utterback T, Watthey L, McDonald L, Artiach P, Bowman C, Garland S, Fuji C, Cotton MD, Horst K, Roberts K, Hatch B, Smith HO, Venter JC. Genomic sequence of a Lyme disease spirochaete, Borrelia burgdorferi. Nature. 1997 Dec 11;390(6660):580-6. doi: 10.1038/37551. PMID 9403685
- [Background] Casjens S, Palmer N, van Vugt R, Huang WM, Stevenson B, Rosa P, Lathigra R, Sutton G, Peterson J, Dodson RJ, Haft D, Hickey E, Gwinn M, White O, Fraser CM. A bacterial genome in flux: the twelve linear and nine circular extrachromosomal DNAs in an infectious isolate of the Lyme disease spirochete Borrelia burgdorferi. Mol Microbiol. 2000 Feb;35(3):490-516. doi: 10.1046/j.1365-2958.2000.01698.x. PMID 10672174